CLINICAL TRIAL: NCT04436536
Title: Gait Speeds and Demands in Chronic Stroke Patients: A Multi-dimensional Investigation
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng Kung University (Other)
Collaborators: Tainan Hospital, Ministry of Health and Welfare (Other)
Responsible Party: Principal Investigator, Sang-I Lin, Professor, Department of Physical Therapy, National Cheng Kung University, National Cheng Kung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-BR-107-101-T
Record Dates: First submitted 2020-06-15; First posted 2020-06-18 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Stroke
Keywords: stroke; gait; dual tasks; motor learning
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- training with random speed changes (Experimental): Walking training on treadmill with random speed changes, that is, random sequence of several different walking speeds
  Interventions: Other: Treadmill walking training with random speed changes
- training with blocked speed changes (Active Comparator): Walking training on treadmill with blocked speed changes, that is a steady progression of faster walking speed.
  Interventions: Other: Treadmill walking training with blocked speed changes

INTERVENTIONS:
Other: Treadmill walking training with random speed changes — Participants were asked to walk in different gait speed randomly on the treadmill (80%, 90%, 100%, 110% and 120% of preferred speed). The training speed would be changed in every 15 seconds in 2-minutes-section. 2 minutes/ section, 10 sections/ day, 3 days/ week, 2 weeks. 1 minute rest time would be held between sections.
  Arms: training with random speed changes
Other: Treadmill walking training with blocked speed changes — Participants were asked to walk in same gait speed on the treadmill per day (80%, 90%, 100%, 110% and 120% of preferred speed, respectively). 2 minutes/ section, 10 sections/ day, 3 days/ week, 2 weeks. 1 minute rest time would be held between sections.
  Arms: training with blocked speed changes

SUMMARY:
This study investigated the effect of treadmill walking training with and without random speed changes in persons in the chronic stage of stroke. It was hypothesized that random speed change group will show less attention and balance demands for speed change in level walking.

DETAILED DESCRIPTION:
This study includes chronic stroke patients who will be randomly assigned to blocked or random walking speed change group to receive 30 min per session, 3 sessions per week for 2 weeks' walking training on a treadmill. The outcome measures include gait characteristics under 3 tasks x 3 speed conditions x 2 attention conditions on an obstacle-free walk way. The three tasks are normal walking, narrow based walking and obstacle crossing. The three speed conditions are constant (preferred) speed, speeding up (preferred to maximum speed), and slowing down (maximum to preferred speed). The two attention conditions are none and serial subtraction of 3 during walking. Clinical sensorimotor function assessment, including hand grip strength, plantar sensitivity, stroke rehabilitation assessment of movement and Fugl-Meyer lower extremity motor scale will be conducted for subject characterization.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with first stroke for at least 6 months
* Able to walk for at least 20 minutes independently without exhaustion
* Residual gait deficits
* Resting blood pressure is lower than 150/90 mmHg

Exclusion Criteria:

* Unable to follow experimental instructions during the process
* Any pain, inflammation, or other neuromuscular or musculoskeletal conditions in the lower limbs that affect walking ability
* Unstable health problems

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-02-26 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
stride characteristics | 2 weeks
  Wearable movement sensors are used to measure stride characteristics, such step length, gait velocity, under different walking conditions (normal, narrow based, dual task)

CONTACTS AND LOCATIONS:
Overall Officials: Lin Sang-I, PhD, Study Chair — National Cheng Kung University
Locations (1):
- National Cheng Kung University, Tainan, Taiwan